CLINICAL TRIAL: NCT04039516
Title: Phase II Randomised Trial to Assess Progression of Carcinoid Heart Disease in Patients Treated With Lutathera Therapy Compared to Best Supportive Care.
Brief Title: Carcinoid Heart Disease and Peptide Receptor Radiotargetted Therapy
Acronym: CHARRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 263064
Record Dates: First submitted 2019-07-05; First posted 2019-07-31 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Carcinoid Heart Disease; Carcinoid Syndrome; Carcinoid Tumor
MeSH Terms: conditions — Carcinoid Heart Disease; Serotonin Syndrome; Carcinoid Tumor | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lutathera Treatment Arm (Experimental): • 4x cycles of 7.4 GBq (200mCi) of Lutathera therapy (177Lu-DOTA0-Tyr3-Octreotate) with concomitant amino acids for participants randomised onto the Lutathera therapy arm, every 8 weeks, plus long term somatostatin analogues (SSTA).
  Interventions: Drug: Lutathera
- Best Supportive Care (No Intervention): Somatostatin analogue treatment according to current standard, routine care

INTERVENTIONS:
Drug: Lutathera — A total of 4 infusions of Lutathera to be administered every 8 weeks.
  Arms: Lutathera Treatment Arm

SUMMARY:
Randomised trial to assess progression of carcinoid heart disease in patients treated with Lutathera therapy compared to best supportive care.

DETAILED DESCRIPTION:
This is an open-label, phase II, multicentre, randomised (1:1) clinical trial of an interventional medicinal product. This study will open at 3 centres across the UK. King's College Hospital NHS Foundation Trust will act as the coordinating centre for the study.

In this study, treatment with Lutathera will be compared to treatment with current best supportive care (somatostatin analogues) in patients with inoperable, somatostatin receptor positive, histologically confirmed small bowel NENs and these patients should have stable disease according to RECIST criteria for a period of 6 months prior to study entry.

Patients on the treatment arm will receive four administrations of 7.4 GBq (200 mCi) of Lutathera (and concomitant amino acids will be given with each administration for kidney protection). Patients are scheduled to continue to receive study treatment until any of the following occurs:

1. Unacceptable toxicity;
2. Progressive disease as determined by RECIST Criteria;
3. Inability or unwillingness of the patient to comply with study procedures;
4. Patient withdraws consent to participate Patients on the best supportive care arm will receive somatostatin analogue treatment every 4 weeks according to local standard of care practices.

Tumour response in both arms will be assessed after cycles 2 and 4 of 177Lu-Dotatate therapy, or every 16 weeks for patients enrolled under the best supportive care arm, according to RECIST criteria.

The study population is comprised of patients with stable carcinoid heart disease (CHD) and carcinoid syndrome. King's College Hospital performed surgery on 30 patients with carcinoid heart disease over the last 5 years. On review of patient records at King's, a further 30 patients with carcinoid heart disease were identified during the same time period who did not require surgery.

Other centres participating in this study have similar populations of patients with CHD, with specific multi-disciplinary team meetings and outpatient clinics for identification and recruitment of suitable patients into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Echocardiographic evidence of mild/ moderate carcinoid heart disease.
2. Carcinoid syndrome with Echocardiographic evidence of carcinoid heart disease- to be defined further
3. Elevated urinary 5-HIAA or NYHA class I or II on therapy [not necessarily exceeding label dose of SSA LAR; eg, could be 30mg SMS LAR plus sc SMS for breakthrough]
4. Presence of metastasized or locally advanced, inoperable (curative intent) histologically proven, Grade 1 or Grade 2 gastroenteropancreatic neuroendocrine (GEP-NET) or Lung-NET tumor
5. Age >18
6. Ki67 index ≤ 20%
7. Patients who have provided a signed informed consent form to participate in the study, obtained prior to the start of any protocol related activities
8. Confirmed presence of somatostatin receptors on all target lesions documented by CT/MRI scans, within 8 weeks prior to randomization (centrally confirmed), as assessed by the following somatostatin receptor imaging (SRI) modalities: [68Ga]-DOTA-TOC (Somakit-TOC™) PET/CT imaging or [68Ga]-DOTA-TATE PET/CT imaging (NETSPOTTM) or Somatostatin Receptor scintigraphy (SRS) with 111In-pentetreotide (Octreoscan®).

10. Irresectable disease 11. Karnofsky Performance Score (KPS) ≥60.

Exclusion Criteria:

1. Patients with progressive disease by RECIST progressed within 6 months
2. Unable to consent
3. Pregnant
4. Chemotherapy within 3 months
5. PRRT within 3 years
6. Grade 3 tumours (WHO 2010)
7. Severe or Uncontrolled carcinoid heart disease
8. Renal impairment with eGRF <40 ml/min
9. NYHA class III,IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The rate of progression of moderate carcinoid heart disease (CHD) | 5 years
  The rate of progression of carcinoid heart disease (CHD) in patients with moderate CHD will be compared across the Lutathera Therapy and Best Supportive Care Arms and will be assessed through RECIST CT/MRI imaging and urinary 5-HIAA levels throughout the duration of the study.
  The rate of progression will be assessed at each study visit across both arms during the intervention and follow-up phase. If the study treatment is successful in delaying the rate of progression, then the rate of progression in the Lutathera (study intervention) arm is expected to be much slower than in the Best Supportive Care arm.

SECONDARY OUTCOMES:
Change in NYHA heart failure score | 5 years
  The association between Lutathera Therapy against Best Supportive Care will be assessed by comparing the change in NYHA heart failure score in patients enrolled in both study arms.
  The NYHA Heart Failure Score is grade I to IV, with Grade I being No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath) and Grade IV being Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  The change in grade will be assessed with an anticipated reduction in grade if the study treatment is successful in reducing symptoms.
Progressive disease | 5 years
  Progressive disease will be determined according to RECIST 2.0 criteria, following imaging (CT/MRI) conducted throughout the study, on all enrolled participants across the Lutathera Therapy and Best Supportive Care arm.
  Tumour size according to RECIST 2.0 criteria will be examined with an anticipated decrease in tumour size should the study intervention be successful.
Reduction in urinary 5-HIAA levels | 5 years
  Reduction in urinary 5-HIAA levels throughout the course of the study will be compared across the Lutathera Therapy and Best Supportive Care arms.
  Elevated 5-HIAA levels are an indicator of Carcinoid Syndrome, which is the condition under study in this clinical trial. A reduction in urinary 5-HIAA levels is expected should the study intervention prove successful.
Change in quality of life measurements (European Organization for Research and Treatment of Cancer questionnaires, QLQ-C30 and QLQ-GI.NET2) | 5 years
  All enrolled patients will be required to complete the following validated quality of life questionnaires:
  - European Organization for Research and Treatment of Cancer questionnaires, QLQ-C30 and QLQ-GI.NET2
  The change in quality of life scores will be compared across the Lutathera Therapy arm and Best Supportive Care arm. If the study intervention is successful in moderating disease, a positive increase in the quality of life scores is expected.

IPD SHARING:
Plan to Share IPD: No
No IPD to be shared with other researchers.